CLINICAL TRIAL: NCT06867549
Title: Slow Wave Induction by Propofol to Eliminate Depression (SWIPED) Stage II
Acronym: SWIPED II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ben J.A. Palanca, Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 202411168; U01MH128483 (NIH)
Record Dates: First submitted 2025-02-25; First posted 2025-03-10 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Propofol; Anesthetics; Electroencephalography

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol infusion -moderate dose (Experimental): Serial propofol infusions to maximally and safely induce unconsciousness and EEG slow waves while minimizing burst suppression. Target brain effect-site concentrations >2.5 mcg/ml. This will be paired with BBTI.
  Interventions: Drug: Propofol; Diagnostic Test: Electroencephalography (EEG); Behavioral: Brief Behavioral Therapy for Insomnia
- Propofol infusion - low dose (Active Comparator): Serial propofol infusions to safely induce unconsciousness while minimizing EEG slow waves and burst suppression.Target brain effect-site concentration of 1-2 mcg/ml. This will be paired with BBTI.
  Interventions: Drug: Propofol; Diagnostic Test: Electroencephalography (EEG); Behavioral: Brief Behavioral Therapy for Insomnia

INTERVENTIONS:
Drug: Propofol — Targeted propofol infusion in TRD patients will induce sedation. Dosage of propofol is determined based upon EEG markers and treatment arm.
  Other Names: anesthetic
Diagnostic Test: Electroencephalography (EEG) — EEG will be recorded during propofol infusion and during overnight sleep. Sleep EEG data will be acquired for a minimum of one night prior to the first sedation session, providing a baseline measure. Additional overnight sleep recordings will be performed on day of sedation and subsequent nights.
Behavioral: Brief Behavioral Therapy for Insomnia — Trained staff will provide evaluation and up to 3 follow up appointments of BBTI for all participants. These will be done remotely to assess behavioral approaches to improve overall sleep habits.
  Other Names: BBTI

SUMMARY:
The investigators hypothesize that brief behavioral therapy and targeted propofol infusion in depressed geriatric patients will augment subsequent slow wave sleep and improve clinical and cognitive outcomes. The team will recruit 70 participants for a double-blinded placebo controlled randomized controlled trial. Two propofol infusions, 2-6 days apart, will be administered, targeting either a low propofol dose arm (minimal EEG slow waves, brain effect-site concentration 1-2 mcg/ml) or moderate dose propofol arm (maximal induction of EEG slow waves, brain effect site concentration of >2.5 mcg/ml). The pharmacologic intervention will be paired with 3-4 sessions of Brief Behavioral Therapy for Insomnia for all participants. To minimize bias, there will be no specific gender or ethnic background consideration for enrollment. This will be a single site investigation at Washington University Medical Center.

DETAILED DESCRIPTION:
Depression in older adults is a leading cause of disability, excess mortality from suicide, and dementia. Cognitive problems and sleep disturbances are common, contributing to recurrence and poor long-term outcomes. Disrupted slow-wave sleep is at the nexus of depression and cognitive dysfunction in older adults. Novel approaches to target this core pathophysiology are lacking. This mechanistic project is designed to elucidate the relationships between TRD and sleep disturbances in older adults. Through personalized infusions targeting electroencephalographic (EEG) patterns, the investigators aim for a systematic characterization of the relationships between the propofol (dose and EEG measures) and enhancement of slow wave sleep, with associated secondary clinical and cognitive outcomes. Through the re-purposing of propofol as a therapeutic probe, this innovative proposal will establish whether EEG slow waves are a viable therapeutic target for novel antidepressant approaches.

Two BBTI sessions will be administered before the propofol infusions, with two additional sessions within 6 weeks after the 2nd infusion. The sessions will completed remotely or in person.

Propofol will be infused through a peripheral IV, with the assistance of target-controlled infusion software and pumps, with an anticipated infusion duration of 2 hours. Concurrent high-density EEG will be acquired. Participants will be discharged home after nurse monitoring and fulfillment of post-anesthetic care unit criteria.

Patients will be instructed by staff on the operation of the SOMNOmedics HST for at-home overnight sleep EEG recordings. Patients will demonstrate the ability to successfully wear the device and initiate recordings without assistance. The device, charger, tablet, and instructional materials will be provided to patients.

Overnight sleep recordings will be obtained prior to the first propofol infusion and on evenings of propofol infusions. Additionally, recordings will be obtained for up to 6 weeks after the final infusion, to evaluate persistence of restoration of sleep architecture.

Primary endpoints will be analyzed based on age, sex, time separating propofol infusions, induction of EEG measures during infusions, pharmacokinetic exposure times at varying concentrations, adherence to BBTI, and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age 60 or greater
* English speaking (as an interpreter will not be readily available should a participant need to convey any safety concerns during the propofol infusion sessions or require guidance on conducting at-home sleep recordings)
* Depression (non-responsive to at least one adequate trial of oral antidepressants for current episode).

Exclusion Criteria:

* Presence of symptomatic coronary artery disease
* Presence of marked congestive heart failure/cardiomyopathy(NYHA > Class III, LVEF <40%, greater than mild RV systolic dysfunction)
* Prior reaction to propofol
* Resting heart rate < 50 bpm
* Treatment with Electroconvulsive therapy/Transcranial Magnetic Stimulation/vagal nerve stimulation within 6 weeks
* Body mass index > 35
* C-SSRS of 4 or greater (active suicidal ideation with some intent and with/without a specific plan)
* MoCA score < 23 (at least mild dementia)
* Schizophrenia
* Bipolar disorder
* Non-prescribed use of amphetamines, opioids, cocaine, or phencyclidine; Urine THC > 150 ng/ml
* Intake of > 14 beers/week (or equivalent)
* Anesthetic exposure in the past 4 weeks
* Concurrent use of benzodiazepines > 2 mg/day lorazepam or equivalent, trazodone > 50 mg/day, or gabapentin > 600mg/day.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in SWS duration | Pre-infusion and on the nights of propofol infusions
  This is the total duration of N3 averaged across infusion nights relative to baseline average. The average change in total duration of N3 infusion nights relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Palanca, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be released in manuscript form. Outcome data will be uploaded to the NIMH Data Archive on a rolling basis. EEG data will be shared via the National Sleep Research Resource within three years of study completion.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within three years of study completion.
Access Criteria: Data use agreements may be required